CLINICAL TRIAL: NCT01117272
Title: Relationship of Metabolic Parameters, Endocrine and Prolactin Levels in Taiwan's Women With Polycystic Ovary Syndrome and Hyperprolactinemia.
Brief Title: The Relationship of PRL and Polycystic Ovary Syndrome (PCOS) in Taiwan's Women
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-98009
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; hyperprolactinemia; obesity; hyperandrogenic
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperprolactinemia; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PCOS group: Who met the 2003 Rotterdam criteria.
- Mild hyperprolactinaemia group: Who were diagnosed with prolactin levels above the upper limit of normal (24.29 ng/ml) and under 100 ng/ml.
- Control group: Without PCOS and with normal prolactin levels.

SUMMARY:
Polycystic ovarian syndrome (PCOS) is the most common endocrine disorder of reproductive-age women. According to Rotterdam 2003 criteria: at least two of three criteria are met, hyperandrogenism, chronic anovulation, and polycystic ovary. PCOS will cause irregular menstrual cycle, infertility, acne, hirsutism, obesity, or/and metabolic syndrome, diabetes that may increase risk of cardiovascular disease.

Hyperprolactinaemia is also a common problem in reproductive aged women. Both hyperprolactinaemia and PCOS had endocrine disorder and irregular menstrual cycle. Investigators hope to collect clinical data from PCOS and prolactinemia patients followed in Wang Fang hospital for many years in endocrinological and metabolical aspects for comparison. Investigators at the same time would like to understand more about other similarities and differences between these two endocrinological dysfunction for future study.

ELIGIBILITY:
Inclusion Criteria:

* PCOM by ultrasound Diagnosis
* Anovulation, Oligo menses
* Hyperandrogenism

Exclusion Criteria:

* Women who had been diagnosed with other etiology that should be excluded in PCOS diagnosis, such as hyperprolactinemia, hypogonadotropic hypogonadism, premature ovarian failure, congenital adrenal hyperplastic, androgen-secreting tumor, Cushing's syndrome, disorders of uterus( such as Asherman's syndrome, Mullerian agenesis), chromosomal anomalies( such as Turner syndrome).
* Women who did not have sufficient clinical or biochemical records.
* Girls who had menarche at <3 years of age and women who were >40 years of age.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Polycystic Ovary syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
hyperprolactin | Who visited the Reproductive Endocrinology Clinic at Taipei Medical University-Wan Fang Medical Center from April 2004 to June 2007

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan